CLINICAL TRIAL: NCT04159116
Title: Development of a Protocol for Prevention and Treatment of Laryngospasm and Other Causes of Hypoxemia Based on Identified Risk Factors in Adult Outpatients Undergoing Esophagogastroduodenoscopy (EGD) Under Monitored Anesthesia Care (MAC)
Brief Title: Prevention and Treatment of Laryngospasm and Hypoxemia Based on Risk Factors in Adult Outpatients Undergoing EGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Envision Healthcare Scientific Intelligence, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRE2019-EGD01
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Laryngospasm; Hypoxemia
MeSH Terms: conditions — Laryngismus; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suctioned Prior to Endoscope (Experimental): This group will be suctioned prophylactically after sedation but prior to introduction of endoscope.
  Interventions: Other: Prophylactic suctioning when clinically indicated
- Standard of Care (Other): This group will be suctioned by anesthesia providers when clinically indicated by copious secretions, coughing, choking or desaturation.
  Interventions: Other: Prophylactic suctioning when clinically indicated

INTERVENTIONS:
Other: Prophylactic suctioning when clinically indicated — Suctioned prophylactically when clinically indicated by copious secretions, coughing, choking or desaturatation

SUMMARY:
The purpose of this study is to identify patient and provider-chosen factors that put patients at risk for the development of hypoxemia (oxygen saturation < 90% for 5 seconds) during endoscopy and to use this knowledge to develop a treatment protocol for specific causes of hypoxemia in adult esophagogastroduodenoscopy outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years
* English speaking
* Mentally competent to sign their own consent for treatment

Exclusion Criteria:

* Poor incisor teeth stability
* Anticipated procedure of greater than 30 minutes
* History of facial or oral surgery and a baseline oxygen saturation of less than 95% on room air

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
Incidence of laryngospasm during EGDs | 2 hours
  Determine if prophylactic suctioning after sedation but prior to introduction of endoscope changes the incidence of laryngospasm during EGDs.
Identify risk factors for the development of hypoxemia during EGD | 2 hours
  These risk factors include both patient factors (ASA class, history of cardiopulmonary disease, BMI, social history, Obstructive Sleep Apnea, STOP-BANG scores and age) and provider-chosen factors (medications given, airway interventions, percent and flow of oxygen in liters per minute, and whether or not the patient was suctioned prior to or during the procedure).

SECONDARY OUTCOMES:
Incidence of copious secretions, choking, desaturation, and shortened or aborted procedures | 2 hours
  Determine if prophylactic suctioning after sedation but prior to introduction of endoscope changes the incidence of copious secretions, choking, desaturation, and shortened or aborted procedures.
Identify the various causes of hypoxemia during EGD | 2 hours
  These risk include apnea, hypoventilation, laryngospasm, or other cause of airway obstruction

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morrison, DNP, CRNA, Principal Investigator — Envision Healthcare
Locations (1):
- Three Rivers Endoscopy, Moon Township, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No